CLINICAL TRIAL: NCT05061797
Title: A Double-Blind, Randomized, Crossover Study to Examine the Thermogenic Effect of an Energy Drink in Healthy Adults
Brief Title: A Study to Examine the Effect of a Thermogenic Energy Drink in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowdy Energy (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Energy Drink in HealthBIO-2113
Record Dates: First submitted 2021-08-30; First posted 2021-09-30 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Metabolism
Keywords: Thermogenic

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Crossover Study
Who Masked: Participant, Investigator
Masking Description: Samples are coded with 3 digit, randomized codes. Active study product and placebo are not known to the administrators of the study or the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Study Product (Active Comparator): An energy beverage formulated to improve the thermogenic (calorie burning) impact in humans via caffeine and ingredients for overall metabolic wellness.
  Interventions: Dietary Supplement: Thermogenic Energy Drink - Active Study Product Formula
- Placebo (Placebo Comparator): A carbonated soft-drink with the same appearance, aroma, and flavor as the active study product
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Thermogenic Energy Drink - Active Study Product Formula — The Thermogenic Energy Drink is the Active Study Product (ASP). This energy drink formula combines, caffeine, guarana, Vitamins C, B3, B6, B12, Magnesium, Potassium, L-Citrulline, L-Arginine HCl, L-Glutamine, and Chlorogenic Acids from green coffee bean extract. Participants will consume an assigned amount of the beverage (355 ml), under observation. They will be monitored for the following 180 minutes with measurements of respiration for Resting Energy Expenditure (RER) and other metabolic markers as well as satiety via Visual Analog Scale (VAS).
  Other Names: Energy Drink - Rowdy Energy
  Arms: Active Study Product
Dietary Supplement: Placebo — A carbonated soft drink with the same appearance, flavor and aroma as the active study product. Study participants will consume an assigned amount of the beverage (355 ml) under observation. They will then be monitored for the subsequent 180 minutes with measurements for respiration for Resting Energy Expenditure (RER) and other metabolic markers as well as satiety via a Visual Analog Scale (VAS).
  Arms: Placebo

SUMMARY:
This study is intended to examine the acute thermogenic effects of the active study product (energy drink), in healthy adults.

DETAILED DESCRIPTION:
The active study product and a control will be blinded with 3 digit codes. Human subjects will consume the coded products in a randomized manner. Measurements of rest energy expenditure via respiration will be performed throughout a 3 hour time span with controlled intervention an observation. Additional metrics will be gathered relating to benefits and/or side effects. The data gathered will be used to calculate the thermogenic impact of the active study product on healthy adults. The study is designed based on statistical confidence, with a minimum required number of active participants set to 26. 30 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy male or female, 18-50 years of age, inclusive.

* BMI of ≥18.0 and ≤30.0 kg/m2 at Visit 1 (Day -7).
* Non-user of all tobacco, smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes), and nicotine products (e.g., nicotine gum and/or nicotine patches) within 1 y of Visit 1 (Day -7) and has no plans to change status during the study period.
* Willing to maintain habitual diet and physical activity patterns throughout the trial.
* Willing and able to comply with the visit schedule.
* Willing to refrain from exclusionary medications, supplements, and products.
* No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator

Exclusion Criteria:

* Known allergy, intolerance, or sensitivity to any of the ingredients in the study product provided.
* Abnormal laboratory test results of clinical significance at Visit 1 (Day -7) at the discretion of the Clinical Investigator. One re-test will be allowed on a separate day prior to Visit 2 (Day 0), for subjects with abnormal laboratory test results.
* Use of hemp or marijuana products within 1 mo of Visit 1 (Day -7)
* Extreme dietary habits at the discretion of the Clinical Investigator.
* Currently or planning to be on a weight loss regimen during the study or use of weight-loss drugs (including over-the-counter medications and/or supplements, including thermogenic/fat-burning supplements) or participated in weight-loss programs within 3 mo of Visit 1 (Day -7).
* Chronic use of products that may affect metabolism (e.g., ephedrine alkaloids, guggulsterones, etc.) and/or muscle mass (i.e. creatine, protein/amino acids (including free and/or branched chain amino acid), androstenedione, dihydroepiandrosterone (DHEA), hydroxylmethylbutyrate, pre/post-workout supplements, etc.) within 3 mo of Visit 1 (Day -7). Non-chronic users (<3 serving/week) must have a 2-wk washout prior to Visit 2 (Day 0).
* History or presence of clinically important endocrine (including hyper/hypo-parathyroidism, type 1 or 2 diabetes mellitus and/or hypoglycemia), cardiovascular (unstable angina pectoris or myocardial infarction, heart failure or cardiomyopathy (acute or chronic), coronary artery revascularization (PCI) or bypass surgery, malignant atrial or ventricular arrhythmia, valvular heart disease or congenital heart disease), pulmonary (including uncontrolled asthma), hepatic, renal (including chronic kidney disease), hematologic (including chronic anemia), immunologic, dermatologic, neurologic, rheumatic (including gout), biliary, polycystic ovarian syndrome, muscle diseases, and/or psychiatric disorders, that, in the opinion of the Clinical Investigator, could interfere with the interpretation of the study results.
* Hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -7). One re-test will be allowed on a separate day prior to Visit 2 (Day 0), for subjects whose blood pressure exceeds either of these cut points at Visit 1 (Day -7), in the judgment of the Clinical Investigator.
* Reports any clinically important gastrointestinal condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, short bowel syndrome, gastroparesis, celiac disease, intestinal dysmotility, active diverticulitis, or ischemic colitis, or any other related condition and subjects with uncontrolled severe diarrhea, nausea or vomiting from any cause, and history of surgery for weight loss), that, in the judgment of the Clinical Investigator, may have the potential to disrupt normal digestion and absorption.
* History or presence of cancer within 5 y of screening (Visit 1, Day -7), except for localized basal cell carcinoma and squamous cell carcinoma of the skin.
* History of active tuberculosis, HIV, AIDS, or Hepatitis-A, -B, and -C.
* Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
* Recent history of (within 12 mo of screening; Visit 1; Day -7) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Exposure to any non-registered drug product within 30 d of Visit 1 (Day -7).
* Use of oral and intravenous antibiotics, antifungals, and antiparasitics within 3 mo of Visit 1 (Day -7). Topical use of antibiotics, antifungals, and antiparasitics will be at the discretion of the Clinical Investigator.
* Unstable use of birth control pills, intrauterine device, and vaginal rings within 3 mo of Visit1 (Day -7).
* Unstable use of inhaled steroids for asthma within 3 mo of Visit 1 (Day -7).
* Regular (daily) use of NSAIDs within 1 mo of Visit 1 (Day -7).
* Use of topical, optical or oral steroids within 1 mo of Visit 1 (Day -7).
* Use of medications known to affect hormones (including, but not limited to progestational agents, estrogen or estrogen receptor modulators, and growth hormone) within 1 mo of Visit1 (Day -7).
* Use of dronabinol within 1 mo of Visit 1 (Day -7).
* Use of metformin within 1 mo of Visit 1 (Day -7).
* Use of prescription strength anti-inflammatories within 48 h of Visit 1 (Day -1).
* Has a condition the Clinical Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Target at least 50% of the participants as "Female." The balance would be male.
Enrollment: 30 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Thermogenic Effect through REE (Resting Energy Expenditure) | Up to 12 weeks for all participants, 180 minutes per participant per session.
  The quantified Thermogenic Impact of the ASP as measured from Resting Energy Expenditure testing with human participants following consumption of the ASP Thermogenic Energy Beverage. This is done via the difference in the net-incremental area under the curve (AUC) for the ASP Thermogenic Beverage vs. the Placebo. A larger difference in REE between the ASP Thermogenic Beverage and the Placebo indicates a greater Thermogenic (calorie expending) effect from the ASP Thermogenic Beverage.

SECONDARY OUTCOMES:
Satiety (As Perceived by the Participant) | Up to 12 weeks for all participants, 180 minutes per participant per session.
  A qualitative review of satiety experienced by study participants using a Visual Analog Scale (VAS). The VAS is measured on a scale of 0 to 100, where 0 indicates no appetite and increasing values indicating higher appetite sensations. The VAS is designed to have participants assess their hunger, desire to eat, and fullness during the 180 minute time span of the test. Lower numerical scores for appetite would indicate improved satiety.
Side Effects/ Gastrointestinal Tolerance | Up to 12 weeks for all participants, 180 minutes per participant per session.
  A qualitative assessment of GI (Gastrointestinal Tolerance) The Participants will complete a Gastrointestinal Tolerance Questionnaire where they will asses and evaluate their symptoms on a scale from 0 to 3, with 0 indicating no experience of the symptom and 3 indicating a severe experience of the symptom. These will include Gat/flatulence, Abdominal Bloating, Abdominal Pain/ Discomfort, Borborygmus/ stomach rumbling, Burping, Reflux, Nausea, Vomiting. Lower scores for all symptoms would indicate that the Thermogenic Energy Drink ASP is well-tolerated.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Chen, Study Director — BioFortis
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amaro-Gahete FJ, Jurado-Fasoli L, De-la-O A, Gutierrez A, Castillo MJ, Ruiz JR. Accuracy and Validity of Resting Energy Expenditure Predictive Equations in Middle-Aged Adults. Nutrients. 2018 Nov 2;10(11):1635. doi: 10.3390/nu10111635. PMID 30400196
- [Background] Bracco D, Ferrarra JM, Arnaud MJ, Jequier E, Schutz Y. Effects of caffeine on energy metabolism, heart rate, and methylxanthine metabolism in lean and obese women. Am J Physiol. 1995 Oct;269(4 Pt 1):E671-8. doi: 10.1152/ajpendo.1995.269.4.E671. PMID 7485480
- [Background] Clark NW, Wells AJ, Coker NA, Goldstein ER, Herring CH, Starling-Smith TM, Varanoske AN, Panissa VLG, Stout JR, Fukuda DH. The acute effects of thermogenic fitness drink formulas containing 140 mg and 100 mg of caffeine on energy expenditure and fat metabolism at rest and during exercise. J Int Soc Sports Nutr. 2020 Feb 13;17(1):10. doi: 10.1186/s12970-020-0341-4. PMID 32054486
- [Background] Compher C, Frankenfield D, Keim N, Roth-Yousey L; Evidence Analysis Working Group. Best practice methods to apply to measurement of resting metabolic rate in adults: a systematic review. J Am Diet Assoc. 2006 Jun;106(6):881-903. doi: 10.1016/j.jada.2006.02.009. PMID 16720129
- [Background] Dulloo AG, Geissler CA, Horton T, Collins A, Miller DS. Normal caffeine consumption: influence on thermogenesis and daily energy expenditure in lean and postobese human volunteers. Am J Clin Nutr. 1989 Jan;49(1):44-50. doi: 10.1093/ajcn/49.1.44. PMID 2912010
- [Background] Fullmer S, Benson-Davies S, Earthman CP, Frankenfield DC, Gradwell E, Lee PS, Piemonte T, Trabulsi J. Evidence analysis library review of best practices for performing indirect calorimetry in healthy and non-critically ill individuals. J Acad Nutr Diet. 2015 Sep;115(9):1417-1446.e2. doi: 10.1016/j.jand.2015.04.003. Epub 2015 May 30. PMID 26038298
- [Background] Thom E. The effect of chlorogenic acid enriched coffee on glucose absorption in healthy volunteers and its effect on body mass when used long-term in overweight and obese people. J Int Med Res. 2007 Nov-Dec;35(6):900-8. doi: 10.1177/147323000703500620. PMID 18035001